CLINICAL TRIAL: NCT01338870
Title: A 12-week, Phase 2, Randomized, Double-blind, Placebo Controlled, Dose-ranging, Parallel Group Study to Evaluate the Efficacy and Safety of Twice Daily Pf-04991532 and Once Daily Sitagliptin in Adult Patients With Type 2 Diabetes Mellitus Inadequately Controlled on Metformin
Brief Title: Study of Safety and Efficacy of PF-04991532 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B2611003
Record Dates: First submitted 2011-04-13; First posted 2011-04-20 (Estimated); Results first posted 2013-04-23 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Phase 2; safety and efficacy study with PF-04991532; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 6-(3-cyclopentyl-2-(4-(trifluoromethyl)-1H-imidazol-1-yl)propanamido)nicotinic acid; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo (Placebo Comparator): Placebo for PF-04991532 and sitagliptin
  Interventions: Drug: Placebo
- 25 mg PF-04991532 (Experimental)
  Interventions: Drug: 25 mg PF-04991532
- 75 mg PF-04991532 (Experimental)
  Interventions: Drug: 75 mg PF-04991532
- 150 mg PF-04991532 (Experimental)
  Interventions: Drug: 150 mg PF-04991532
- 300 mg PF-04991532 (Experimental)
  Interventions: Drug: 300 mg PF-04991532
- Sitagliptin 100 mg (Active Comparator)
  Interventions: Drug: Sitagliptin 100 mg

INTERVENTIONS:
Drug: Placebo — Tablets (n=4), 0 mg twice daily for 84 days
  Arms: Placebo
Drug: 25 mg PF-04991532 — Tablets (n=1), 25 mg strength + tablets (n=3) 0 mg twice daily for 84 days
  Arms: 25 mg PF-04991532
Drug: 75 mg PF-04991532 — Tablets (n=3), 25 mg strength + tablets (n=1) 0 mg twice daily for 84 days
  Arms: 75 mg PF-04991532
Drug: 150 mg PF-04991532 — Tablets (n=1), 150 mg strength + tablets (n=3) 0 mg twice daily for 84 days
  Arms: 150 mg PF-04991532
Drug: 300 mg PF-04991532 — Tablets (n=2), 150 mg strength + tablets (n=2) 0 mg twice daily for 84 days
  Arms: 300 mg PF-04991532
Drug: Sitagliptin 100 mg — Tablets (n=1), 100 mg strength + tablets (n=3) 0 mg once daily in the morning for 84 days; and tablets (n=4) 0 mg once daily in the evening for 84 days.
  Arms: Sitagliptin 100 mg

SUMMARY:
B2611003 is designed to study how safe and effective an investigational medication (PF-04991532) is in people with Type 2 diabetes. Subjects in the study will receive 1 of 6 treatments for 3 months. One of the treatments will be sitagliptin which is an approved drug, and another treatment will be placebo, which does not contain active ingredient.

ELIGIBILITY:
Inclusion Criteria:

Subjects with type 2 diabetes on stable doses of background medicines for management of diabetes; aged 18-70 years; body mass index between 22.5 and 45.5 kg/m2

Exclusion Criteria:

Subjects with type 1 diabetes, heart attack or stroke in the past 6 months, uncontrolled blood pressure, significant kidney disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2011-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (42):
- United States (25):
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Roseville, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Coral Gables, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Augusta, Kansas
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Lake Charles, Louisiana
  - Pfizer Investigational Site, Auburn, Maine
  - Pfizer Investigational Site, Brooklyn Center, Minnesota
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Trenton, New Jersey
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Fargo, North Dakota
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Lansdale, Pennsylvania
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Katy, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
- Canada (6):
  - Pfizer Investigational Site, Surrey, British Columbia
  - Pfizer Investigational Site, Bay Roberts, Newfoundland and Labrador
  - Pfizer Investigational Site, Brampton, Ontario
  - Pfizer Investigational Site, Mississauga, Ontario
  - Pfizer Investigational Site, Mirabel, Quebec
  - Pfizer Investigational Site, Québec, Quebec
- Hungary (2):
  - Pfizer Investigational Site, Balatonfüred
  - Pfizer Investigational Site, Kistelek
- Mexico (3):
  - Pfizer Investigational Site, Aguascalientes, Aguascalientes
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Tlalnepantla, State of Mexico
- Slovakia (4):
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Nové Mesto nad Váhom
  - Pfizer Investigational Site, Pezinok
  - Pfizer Investigational Site, Prešov
- Taiwan (2):
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Taoyuan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2611003&StudyName=Study%20of%20Safety%20and%20Efficacy%20of%20PF-04991532%20in%20Subjects%20with%20Type%202%20Diabetes

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants received placebo matched to PF-04991532 or placebo matched to sitagliptin tablet orally twice daily along with background metformin immediate release tablets, during the 2-week run-in period. Compliant participants were then randomized to study treatments for 12 weeks.
Groups:
- Placebo: Placebo matched to PF-04991532 tablets orally twice daily or placebo matched to sitagliptin tablet orally twice daily along with background metformin 500 milligram (mg) immediate release tablets or as per standard clinical practice (based on the dose prior to randomization), for 12 weeks.
- PF-04991532 25 mg: PF-04991532 25 mg tablet orally twice daily along with background metformin 500 mg immediate release tablets or as per standard clinical practice (based on the dose prior to randomization), for 12 weeks.
- PF-04991532 75 mg: PF-04991532 75 mg tablet orally twice daily along background metformin 500 mg immediate release tablets or as per standard clinical practice (based on the dose prior to randomization), for 12 weeks.
- PF-04991532 150 mg: PF-04991532 150 mg tablet orally twice daily along with background metformin 500 mg immediate release tablets or as per standard clinical practice (based on the dose prior to randomization), for 12 weeks.
- PF-04991532 300 mg: PF-04991532 300 mg tablet orally twice daily along with background metformin 500 mg immediate release tablets or as per standard clinical practice (based on the dose prior to randomization), for 12 weeks.
- Sitagliptin 100 mg: Sitagliptin 100 mg tablet orally once daily as morning dose and placebo matched to sitagliptin tablet orally once daily as evening dose along with background metformin 500 mg immediate release tablets or as per standard clinical practice (based on the dose prior to randomization), for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg | Sitagliptin 100 mg
Started | 50 | 49 | 50 | 50 | 52 | 50
Completed | 41 | 37 | 39 | 41 | 46 | 44
Not Completed | 9 | 12 | 11 | 9 | 6 | 6
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 4 | 0 | 0 | 2
Not completed — Other | 3 | 3 | 3 | 2 | 0 | 2
Not completed — Protocol Violation | 0 | 2 | 2 | 2 | 1 | 1
Not completed — Adverse Event | 4 | 4 | 1 | 5 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg | Sitagliptin 100 mg | Total
Number analyzed (Participants) | 50 | 49 | 50 | 50 | 52 | 50 | 301
Age Continuous [Mean (Standard Deviation); unit: years] | 55.7 (8.8) | 59.2 (6.8) | 56.1 (8.6) | 57.2 (8.7) | 56.0 (7.7) | 55.6 (9.0) | 56.6 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 30 | 21 | 20 | 30 | 15 | 132
  Male | 34 | 19 | 29 | 30 | 22 | 35 | 169

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 12
Description: HbA1c is a form of hemoglobin which is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. The normal range for the HbA1c test is between 4 percent (%) and 5.6%. HbA1c levels between 5.7% and 6.4% indicate increased risk of diabetes and levels of 6.5% or higher indicate diabetes.
Time Frame: Baseline, Week 12
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of study medication. Here 'n' signifies participants who were evaluable at specific time point for each treatment arm respectively.
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin
Arm/Group | Placebo | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 50 | 49 | 50 | 50 | 52 | 50
percentage of hemoglobin
  Baseline (n= 50, 49, 50, 50, 52, 50) | 8.11 (1.255) | 7.90 (0.939) | 7.86 (0.998) | 7.93 (1.018) | 8.01 (1.064) | 8.05 (0.958)
  Change at Week 12 (n= 42, 37, 39, 40, 46, 44) | -0.30 (0.681) | -0.15 (0.593) | -0.51 (0.847) | -0.36 (0.828) | -0.79 (0.743) | -0.65 (0.754)
Statistical Analysis 1: Comparison: Placebo vs PF-04991532 25 mg; Treatment difference and 80% confidence interval (CI) were based on least squares (LS) mean. A mixed model repeated measure (MMRM) analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline, baseline-by-time interaction, baseline-by-treatment interaction, baseline-by-treatment-by-time interaction as the covariates, time was repeated for participant; Test type: Superiority or Other; p = 0.7606, Mixed Models Analysis; Least squares (LS) mean difference = 0.10, 80% CI 2-sided [-0.08 to 0.29], Standard Error of Mean 0.145
Statistical Analysis 2: Comparison: Placebo vs PF-04991532 75 mg; Treatment difference and 80% CI were based on LS mean. A MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline, baseline-by-time interaction, baseline-by-treatment interaction, baseline-by-treatment-by-time interaction as the covariates, time was repeated for participant; Test type: Superiority or Other; p = 0.0266, Mixed Models Analysis; LS mean difference = -0.28, 80% CI 2-sided [-0.46 to -0.09], Standard Error of Mean 0.142
Statistical Analysis 3: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0440, Mixed Models Analysis; LS mean difference = -0.24, 80% CI 2-sided [-0.42 to -0.06], Standard Error of Mean 0.141
Statistical Analysis 4: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; LS mean difference = -0.53, 80% CI 2-sided [-0.71 to -0.36], Standard Error of Mean 0.137
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0013, Mixed Models Analysis; LS mean difference = -0.43, 80% CI 2-sided [-0.60 to -0.25], Standard Error of Mean 0.139

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 1, 2, 4, 8 and 12
Time Frame: Baseline, Week 1, 2, 4, 8, 12
Population: FAS included all randomized participants who received at least 1 dose of study medication. Here 'n' signifies participants who were evaluable at specific time point for each treatment arm respectively.
Measure: Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)
Arm/Group | Placebo | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 50 | 49 | 50 | 50 | 52 | 50
milligram/deciliter (mg/dL)
  Baseline (n= 50, 49, 50, 50 ,52, 50) | 168.41 (51.859) | 167.71 (52.401) | 161.43 (43.009) | 163.38 (44.976) | 168.87 (47.630) | 170.42 (41.366)
  Change at Week 1 (n= 48, 47, 47, 46, 46, 45) | 3.69 (24.632) | -0.70 (26.644) | -3.29 (20.131) | -3.75 (19.486) | -15.35 (35.673) | -18.59 (30.637)
  Change at Week 2 (n= 44, 44, 45, 45, 47, 48) | -1.31 (21.746) | 1.05 (22.186) | -3.84 (24.007) | -1.68 (26.966) | -16.68 (43.620) | -20.13 (32.632)
  Change at Week 4 (n= 46, 42, 44, 45, 48, 49) | 2.00 (36.067) | 6.08 (24.687) | -6.56 (32.880) | 3.61 (36.385) | -19.84 (31.334) | -18.90 (28.434)
  Change at Week 8 (n= 43, 40, 41, 42, 46, 45) | 5.63 (26.183) | 9.42 (28.172) | -4.98 (30.696) | 4.43 (28.491) | -14.24 (42.128) | -17.84 (28.715)
  Change at Week 12 (n= 42, 37, 38, 40, 46, 44) | 3.41 (34.430) | 8.06 (23.298) | -6.55 (31.919) | 6.20 (38.122) | -16.80 (35.765) | -16.07 (31.298)
Statistical Analysis 1: Comparison: Placebo vs PF-04991532 25 mg; Week 1: Treatment difference and 95% CI were based on LS mean. MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.3611, Mixed Models Analysis; LS mean difference = -5.21, 95% CI 2-sided [-16.40 to 5.98], Standard Error of Mean 5.700
Statistical Analysis 2: Comparison: Placebo vs PF-04991532 75 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0969, Mixed Models Analysis; LS mean difference = -9.45, 95% CI 2-sided [-20.61 to 1.71], Standard Error of Mean 5.686
Statistical Analysis 3: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1566, Mixed Models Analysis; LS mean difference = -8.10, 95% CI 2-sided [-19.30 to 3.11], Standard Error of Mean 5.710
Statistical Analysis 4: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0052, Mixed Models Analysis; LS mean difference = -15.92, 95% CI 2-sided [-27.06 to -4.77], Standard Error of Mean 5.678
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; LS mean difference = -21.09, 95% CI 2-sided [-32.30 to -9.88], Standard Error of Mean 5.712
Statistical Analysis 6: Comparison: Placebo vs PF-04991532 25 mg; Week 2: Treatment difference and 95% CI were based on LS mean. MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.9893, Mixed Models Analysis; LS mean difference = 0.08, 95% CI 2-sided [-11.41 to 11.56], Standard Error of Mean 5.852
Statistical Analysis 7: Comparison: Placebo vs PF-04991532 75 mg; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.4767, Mixed Models Analysis; LS mean difference = -4.14, 95% CI 2-sided [-15.55 to 7.27], Standard Error of Mean 5.814
Statistical Analysis 8: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.6222, Mixed Models Analysis; LS mean difference = -2.87, 95% CI 2-sided [-14.28 to 8.55], Standard Error of Mean 5.816
Statistical Analysis 9: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.0159, Mixed Models Analysis; LS mean difference = -13.88, 95% CI 2-sided [-25.16 to -2.61], Standard Error of Mean 5.744
Statistical Analysis 10: Comparison: Placebo vs Sitagliptin 100 mg; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.0012, Mixed Models Analysis; LS mean difference = -18.69, 95% CI 2-sided [-29.95 to -7.44], Standard Error of Mean 5.735
Statistical Analysis 11: Comparison: Placebo vs PF-04991532 25 mg; Week 4: Treatment difference and 95% CI were based on LS mean. MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.5125, Mixed Models Analysis; LS mean difference = 3.86, 95% CI 2-sided [-7.71 to 15.43], Standard Error of Mean 5.895
Statistical Analysis 12: Comparison: Placebo vs PF-04991532 75 mg; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.1455, Mixed Models Analysis; LS mean difference = -8.47, 95% CI 2-sided [-19.89 to 2.94], Standard Error of Mean 5.815
Statistical Analysis 13: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.8712, Mixed Models Analysis; LS mean difference = 0.94, 95% CI 2-sided [-10.43 to 12.31], Standard Error of Mean 5.794
Statistical Analysis 14: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; LS mean difference = -19.57, 95% CI 2-sided [-30.77 to -8.36], Standard Error of Mean 5.707
Statistical Analysis 15: Comparison: Placebo vs Sitagliptin 100 mg; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis; LS mean difference = -19.08, 95% CI 2-sided [-30.26 to -7.90], Standard Error of Mean 5.696
Statistical Analysis 16: Comparison: Placebo vs PF-04991532 25 mg; Week 8: Treatment difference and 95% CI were based on LS mean. MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.2488, Mixed Models Analysis; LS mean difference = 6.99, 95% CI 2-sided [-4.90 to 18.87], Standard Error of Mean 6.055
Statistical Analysis 17: Comparison: Placebo vs PF-04991532 75 mg; [analysis description as in outcome 2, analysis 16]; Test type: Superiority or Other; p = 0.2084, Mixed Models Analysis; LS mean difference = -7.56, 95% CI 2-sided [-19.34 to 4.23], Standard Error of Mean 6.004
Statistical Analysis 18: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 2, analysis 16]; Test type: Superiority or Other; p = 0.9053, Mixed Models Analysis; LS mean difference = 0.71, 95% CI 2-sided [-11.01 to 12.43], Standard Error of Mean 5.971
Statistical Analysis 19: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 2, analysis 16]; Test type: Superiority or Other; p = 0.0091, Mixed Models Analysis; LS mean difference = -15.30, 95% CI 2-sided [-26.79 to -3.81], Standard Error of Mean 5.853
Statistical Analysis 20: Comparison: Placebo vs Sitagliptin 100 mg; [analysis description as in outcome 2, analysis 16]; Test type: Superiority or Other; p = 0.0016, Mixed Models Analysis; LS mean difference = -18.62, 95% CI 2-sided [-30.15 to -7.09], Standard Error of Mean 5.875
Statistical Analysis 21: Comparison: Placebo vs PF-04991532 25 mg; Week 12: Treatment difference and 95% CI were based on LS mean. MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.2963, Mixed Models Analysis; LS mean difference = 6.50, 95% CI 2-sided [-5.71 to 18.70], Standard Error of Mean 6.217
Statistical Analysis 22: Comparison: Placebo vs PF-04991532 75 mg; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.1159, Mixed Models Analysis; LS mean difference = -9.71, 95% CI 2-sided [-21.82 to 2.40], Standard Error of Mean 6.170
Statistical Analysis 23: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.4413, Mixed Models Analysis; LS mean difference = 4.70, 95% CI 2-sided [-7.28 to 16.68], Standard Error of Mean 6.103
Statistical Analysis 24: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.0099, Mixed Models Analysis; LS mean difference = -15.30, 95% CI 2-sided [-26.91 to -3.68], Standard Error of Mean 5.918
Statistical Analysis 25: Comparison: Placebo vs Sitagliptin 100 mg; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.0126, Mixed Models Analysis; LS mean difference = -14.95, 95% CI 2-sided [-26.69 to -3.21], Standard Error of Mean 5.981

3. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 1, 2, 4 and 8
Description: HbA1c is a form of hemoglobin which is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. The normal range for the HbA1c test is between 4% and 5.6%. HbA1c levels between 5.7% and 6.4% indicate increased risk of diabetes and levels of 6.5% or higher indicate diabetes.
Time Frame: Baseline, Week 1, 2, 4, 8
Population: FAS included all randomized participants who received at least 1 dose of study medication. Here, N (number of participants analyzed) signify those who were evaluable for this measure and 'n' signifies participants who were evaluable at specific time point for each treatment arm respectively.
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin
Arm/Group | Placebo | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 48 | 47 | 47 | 46 | 48 | 49
percentage of hemoglobin
  Change at Week 1 (n= 48, 47, 47, 46, 46, 47) | 0.03 (0.496) | -0.01 (0.190) | -0.07 (0.182) | -0.06 (0.227) | -0.02 (0.210) | -0.14 (0.223)
  Change at Week 2 (n= 45, 44, 45, 45, 47, 48) | -0.02 (0.481) | -0.10 (0.236) | -0.08 (0.230) | -0.06 (0.342) | -0.17 (0.275) | -0.21 (0.357)
  Change at Week 4 (n= 46, 42, 44, 45, 48, 49) | -0.14 (0.558) | -0.15 (0.326) | -0.26 (0.436) | -0.32 (0.525) | -0.37 (0.395) | -0.40 (0.463)
  Change at Week 8 (n= 43, 40, 41, 42, 45, 45) | -0.26 (0.615) | -0.14 (0.492) | -0.40 (0.697) | -0.42 (0.708) | -0.58 (0.607) | -0.54 (0.696)
Statistical Analysis 1: Comparison: Placebo vs PF-04991532 25 mg; Week 1: Treatment difference and 80% CI were based on LS mean. MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline, baseline-by-time interaction, baseline-by-treatment interaction, baseline-by-treatment-by-time interaction as the covariates, time was repeated for participant; Test type: Superiority or Other; p = 0.1797, Mixed Models Analysis; LS mean difference = -0.05, 80% CI 2-sided [-0.13 to 0.02], Standard Error of Mean 0.058
Statistical Analysis 2: Comparison: Placebo vs PF-04991532 75 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0234, Mixed Models Analysis; LS mean difference = -0.12, 95% CI 2-sided [-0.19 to -0.04], Standard Error of Mean 0.058
Statistical Analysis 3: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0400, Mixed Models Analysis; LS mean difference = -0.10, 80% CI 2-sided [-0.18 to -0.03], Standard Error of Mean 0.058
Statistical Analysis 4: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.1568, Mixed Models Analysis; LS mean difference = -0.06, 80% CI 2-sided [-0.13 to 0.02], Standard Error of Mean 0.057
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0010, Mixed Models Analysis; LS mean difference = -0.18, 80% CI 2-sided [-0.25 to -0.11], Standard Error of Mean 0.058
Statistical Analysis 6: Comparison: Placebo vs PF-04991532 25 mg; Week 2: Treatment difference and 80% CI were based on LS mean. MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline, baseline-by-time interaction, baseline-by-treatment interaction, baseline-by-treatment-by-time interaction as the covariates, time was repeated for participant; Test type: Superiority or Other; p = 0.0695, Mixed Models Analysis; LS mean difference = -0.10, 80% CI 2-sided [-0.19 to -0.01], Standard Error of Mean 0.070
Statistical Analysis 7: Comparison: Placebo vs PF-04991532 75 mg; [analysis description as in outcome 3, analysis 6]; Test type: Superiority or Other; p = 0.0636, Mixed Models Analysis; LS mean difference = -0.11, 80% CI 2-sided [-0.20 to -0.02], Standard Error of Mean 0.069
Statistical Analysis 8: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 3, analysis 6]; Test type: Superiority or Other; p = 0.0512, Mixed Models Analysis; LS mean difference = -0.11, 80% CI 2-sided [-0.20 to -0.02], Standard Error of Mean 0.069
Statistical Analysis 9: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 3, analysis 6]; Test type: Superiority or Other; p = 0.0051, Mixed Models Analysis; LS mean difference = -0.18, 80% CI 2-sided [-0.26 to -0.09], Standard Error of Mean 0.068
Statistical Analysis 10: Comparison: Placebo vs Sitagliptin 100 mg; [analysis description as in outcome 3, analysis 6]; Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis; LS mean difference = -0.22, 80% CI 2-sided [-0.30 to -0.13], Standard Error of Mean 0.069
Statistical Analysis 11: Comparison: Placebo vs PF-04991532 25 mg; Week 4: Treatment difference and 80% CI were based on LS mean. MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline, baseline-by-time interaction, baseline-by-treatment interaction, baseline-by-treatment-by-time interaction as the covariates, time was repeated for participant; Test type: Superiority or Other; p = 0.2392, Mixed Models Analysis; LS mean difference = -0.07, 80% CI 2-sided [-0.19 to 0.05], Standard Error of Mean 0.094
Statistical Analysis 12: Comparison: Placebo vs PF-04991532 75 mg; [analysis description as in outcome 3, analysis 11]; Test type: Superiority or Other; p = 0.0308, Mixed Models Analysis; LS mean difference = -0.17, 80% CI 2-sided [-0.29 to -0.05], Standard Error of Mean 0.091
Statistical Analysis 13: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 3, analysis 11]; Test type: Superiority or Other; p = 0.0019, Mixed Models Analysis; LS mean difference = -0.27, 80% CI 2-sided [-0.38 to -0.15], Standard Error of Mean 0.091
Statistical Analysis 14: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 3, analysis 11]; Test type: Superiority or Other; p = 0.0034, Mixed Models Analysis; LS mean difference = -0.24, 80% CI 2-sided [-0.36 to -0.13], Standard Error of Mean 0.089
Statistical Analysis 15: Comparison: Placebo vs Sitagliptin 100 mg; [analysis description as in outcome 3, analysis 11]; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; LS mean difference = -0.32, 80% CI 2-sided [-0.44 to -0.21], Standard Error of Mean 0.090
Statistical Analysis 16: Comparison: Placebo vs PF-04991532 25 mg; Week 8: Treatment difference and 80% CI were based on LS mean. MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline, baseline-by-time interaction, baseline-by-treatment interaction, baseline-by-treatment-by-time interaction as the covariates, time was repeated for participant; Test type: Superiority or Other; p = 0.7854, Mixed Models Analysis; LS mean difference = 0.10, 80% CI 2-sided [-0.06 to 0.26], Standard Error of Mean 0.126
Statistical Analysis 17: Comparison: Placebo vs PF-04991532 75 mg; [analysis description as in outcome 3, analysis 16]; Test type: Superiority or Other; p = 0.0778, Mixed Models Analysis; LS mean difference = -0.18, 80% CI 2-sided [-0.33 to -0.02], Standard Error of Mean 0.123
Statistical Analysis 18: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 3, analysis 16]; Test type: Superiority or Other; p = 0.0065, Mixed Models Analysis; LS mean difference = -0.31, 80% CI 2-sided [-0.46 to -0.15], Standard Error of Mean 0.122
Statistical Analysis 19: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 3, analysis 16]; Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis; LS mean difference = -0.37, 80% CI 2-sided [-0.52 to -0.21], Standard Error of Mean 0.119
Statistical Analysis 20: Comparison: Placebo vs Sitagliptin 100 mg; [analysis description as in outcome 3, analysis 16]; Test type: Superiority or Other; p = 0.0013, Mixed Models Analysis; LS mean difference = -0.37, 80% CI 2-sided [-0.52 to -0.21], Standard Error of Mean 0.121

4. Secondary Outcome: Percentage of Participants Achieving Less Than (<) 6.5% or <7% Glycosylated Hemoglobin (HbA1c) Levels
Description: HbA1c is a form of hemoglobin which is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. The normal range for the HbA1c test is between 4% and 5.6%. HbA1c levels between 5.7% and 6.4% indicate increased risk of diabetes, and levels of 6.5% or higher indicate diabetes.
Time Frame: Week 12
Population: FAS included all randomized participants who received at least 1 dose of study medication. Here, N (number of participants analyzed) signify those who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 46 | 44
percentage of participants
  < 6.5% | 11.9 | 8.1 | 15.4 | 17.5 | 17.4 | 15.9
  < 7% | 23.8 | 29.7 | 38.5 | 35.0 | 43.5 | 36.4

5. Secondary Outcome: Change From Baseline in Body Weight at Week 1, 2, 4, 8 and 12
Description: Overweight or obesity increases the risk for developing diabetes. The treatment of diabetes has been the recommendation to lose weight. As weight loss progresses and is maintained, an improvement of glycemia may be evidenced by a reduction in HbA1c.
Time Frame: Baseline, Week 1, 2, 4, 8, 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Placebo | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 50 | 49 | 50 | 50 | 52 | 50
kilogram (kg)
  Baseline (n= 50, 49, 50, 50, 52, 50) | 89.69 (17.571) | 87.24 (19.805) | 85.69 (19.805) | 85.44 (18.305) | 91.61 (21.822) | 91.00 (21.013)
  Change at Week 1 (n= 48, 47, 47, 46, 47, 47) | 0.01 (0.792) | -0.20 (1.170) | 0.14 (1.600) | -0.20 (0.861) | -0.20 (1.168) | -0.33 (2.089)
  Change at Week 2 (n= 45, 44, 45, 45, 47, 48) | 0.31 (2.041) | -0.49 (1.462) | 0.07 (1.510) | -0.25 (1.086) | -0.03 (1.414) | -0.32 (2.488)
  Change at Week 4 (n= 46, 42, 44, 45, 48, 49) | -0.10 (1.255) | -0.55 (1.576) | 0.20 (1.594) | -0.27 (1.381) | -0.58 (1.401) | -0.30 (2.276)
  Change at Week 8 (n= 43, 40, 41, 42, 46, 45) | -0.21 (1.848) | -0.57 (1.488) | -0.04 (2.318) | -0.64 (1.538) | -0.67 (1.649) | -0.61 (2.648)
  Change at Week 12 (n= 42, 37, 39, 41, 46, 44) | -0.30 (1.869) | -0.71 (1.980) | -0.15 (2.757) | -0.83 (2.099) | -0.75 (2.087) | -0.83 (3.026)
Statistical Analysis 1: Comparison: Placebo vs PF-04991532 25 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.5636, Mixed Models Analysis; LS mean difference = -0.16, 95% CI 2-sided [-0.69 to 0.38], Standard Error of Mean 0.272
Statistical Analysis 2: Comparison: Placebo vs PF-04991532 75 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.4889, Mixed Models Analysis; LS mean difference = 0.19, 95% CI 2-sided [-0.35 to 0.72], Standard Error of Mean 0.271
Statistical Analysis 3: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.5849, Mixed Models Analysis; LS mean difference = -0.15, 95% CI 2-sided [-0.68 to 0.39], Standard Error of Mean 0.272
Statistical Analysis 4: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.5104, Mixed Models Analysis; LS mean difference = -0.18, 95% CI 2-sided [-0.70 to 0.35], Standard Error of Mean 0.268
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2640, Mixed Models Analysis; LS mean difference = -0.30, 95% CI 2-sided [-0.83 to 0.23], Standard Error of Mean 0.269
Statistical Analysis 6: Comparison: Placebo vs PF-04991532 25 mg; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.0464, Mixed Models Analysis; LS mean difference = -0.71, 95% CI 2-sided [-1.42 to -0.01], Standard Error of Mean 0.357
Statistical Analysis 7: Comparison: Placebo vs PF-04991532 75 mg; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.7107, Mixed Models Analysis; LS mean difference = -0.13, 95% CI 2-sided [-0.83 to 0.56], Standard Error of Mean 0.353
Statistical Analysis 8: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.1564, Mixed Models Analysis; LS mean difference = -0.50, 95% CI 2-sided [-1.19 to 0.19], Standard Error of Mean 0.352
Statistical Analysis 9: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.3834, Mixed Models Analysis; LS mean difference = -0.30, 95% CI 2-sided [-0.98 to 0.38], Standard Error of Mean 0.345
Statistical Analysis 10: Comparison: Placebo vs Sitagliptin 100 mg; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.1279, Mixed Models Analysis; LS mean difference = -0.53, 95% CI 2-sided [-1.21 to 0.15], Standard Error of Mean 0.346
Statistical Analysis 11: Comparison: Placebo vs PF-04991532 25 mg; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.2520, Mixed Models Analysis; LS mean difference = -0.39, 95% CI 2-sided [-1.06 to 0.28], Standard Error of Mean 0.339
Statistical Analysis 12: Comparison: Placebo vs PF-04991532 75 mg; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.2772, Mixed Models Analysis; LS mean difference = 0.37, 95% CI 2-sided [-0.30 to 1.03], Standard Error of Mean 0.336
Statistical Analysis 13: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.7038, Mixed Models Analysis; LS mean difference = -0.13, 95% CI 2-sided [-0.79 to 0.53], Standard Error of Mean 0.335
Statistical Analysis 14: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.2031, Mixed Models Analysis; LS mean difference = -0.42, 95% CI 2-sided [-1.07 to 0.23], Standard Error of Mean 0.329
Statistical Analysis 15: Comparison: Placebo vs Sitagliptin 100 mg; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.6948, Mixed Models Analysis; LS mean difference = -0.13, 95% CI 2-sided [-0.78 to 0.52], Standard Error of Mean 0.330
Statistical Analysis 16: Comparison: Placebo vs PF-04991532 25 mg; [analysis description as in outcome 2, analysis 16]; Test type: Superiority or Other; p = 0.5691, Mixed Models Analysis; LS mean difference = -0.24, 95% CI 2-sided [-1.07 to 0.59], Standard Error of Mean 0.421
Statistical Analysis 17: Comparison: Placebo vs PF-04991532 75 mg; [analysis description as in outcome 2, analysis 16]; Test type: Superiority or Other; p = 0.3447, Mixed Models Analysis; LS mean difference = 0.39, 95% CI 2-sided [-0.42 to 1.21], Standard Error of Mean 0.415
Statistical Analysis 18: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 2, analysis 16]; Test type: Superiority or Other; p = 0.5769, Mixed Models Analysis; LS mean difference = -0.23, 95% CI 2-sided [-1.04 to 0.58], Standard Error of Mean 0.413
Statistical Analysis 19: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 2, analysis 16]; Test type: Superiority or Other; p = 0.3599, Mixed Models Analysis; LS mean difference = -0.37, 95% CI 2-sided [-1.16 to 0.42], Standard Error of Mean 0.402
Statistical Analysis 20: Comparison: Placebo vs Sitagliptin 100 mg; [analysis description as in outcome 2, analysis 16]; Test type: Superiority or Other; p = 0.4600, Mixed Models Analysis; LS mean difference = -0.30, 95% CI 2-sided [-1.10 to 0.50], Standard Error of Mean 0.407
Statistical Analysis 21: Comparison: Placebo vs PF-04991532 25 mg; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.4253, Mixed Models Analysis; LS mean difference = -0.40, 95% CI 2-sided [-1.39 to 0.59], Standard Error of Mean 0.504
Statistical Analysis 22: Comparison: Placebo vs PF-04991532 75 mg; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.4349, Mixed Models Analysis; LS mean difference = 0.39, 95% CI 2-sided [-0.59 to 1.37], Standard Error of Mean 0.497
Statistical Analysis 23: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.6697, Mixed Models Analysis; LS mean difference = -0.21, 95% CI 2-sided [-1.18 to 0.76], Standard Error of Mean 0.492
Statistical Analysis 24: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.5501, Mixed Models Analysis; LS mean difference = -0.28, 95% CI 2-sided [-1.22 to 0.65], Standard Error of Mean 0.476
Statistical Analysis 25: Comparison: Placebo vs Sitagliptin 100 mg; [analysis description as in outcome 2, analysis 21]; Test type: Superiority or Other; p = 0.4081, Mixed Models Analysis; LS mean difference = -0.40, 95% CI 2-sided [-1.35 to 0.55], Standard Error of Mean 0.484

6. Secondary Outcome: Percentage of Participants With Greater Than or Equal to (>=) 1% or >= 2% Gain in Body Weight From Baseline
Description: Overweight or obesity increases the risk for developing diabetes. Participants with >= 1% or >= 2% gain in body weight from baseline signifies a higher risk of diabetes.
Time Frame: Week 12
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 42 | 37 | 39 | 41 | 46 | 44
percentage of participants
  >= 1% | 23.81 | 27.03 | 38.46 | 21.95 | 15.22 | 31.82
  >= 2% | 2.38 | 2.70 | 15.38 | 7.32 | 6.52 | 15.91

7. Secondary Outcome: Percentage of Participants With Greater Than or Equal to (>=) 1% or >= 2% Loss in Body Weight From Baseline
Description: The treatment of diabetes has been the recommendation to lose weight. As weight loss progresses and is maintained, an improvement of glycemia may be evidenced by a reduction in HbA1c. Participants with >= 1% or >= 2% loss in body weight from baseline signifies an improvement of glycemia.
Time Frame: Week 12
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 42 | 37 | 39 | 41 | 46 | 44
percentage of participants
  >= 1% | 38.10 | 35.14 | 30.77 | 48.78 | 41.30 | 40.91
  >= 2% | 23.81 | 27.03 | 17.95 | 26.83 | 30.43 | 29.55

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg | Sitagliptin 100 mg
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/49 | 0/50 | 0/50 | 0/52 | 0/50
Other Adverse Events (participants affected / at risk) | 14/50 | 16/49 | 14/50 | 11/50 | 15/52 | 11/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=50) | PF-04991532 25 mg (N=49) | PF-04991532 75 mg (N=50) | PF-04991532 150 mg (N=50) | PF-04991532 300 mg (N=52) | Sitagliptin 100 mg (N=50)
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 3 | 1 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 4
Pharyngitis (Infections and infestations) | 1 | 2 | 2 | 1 | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 3 | 2 | 2 | 1
Urinary tract infection (Infections and infestations) | 5 | 1 | 2 | 3 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 5 | 0 | 3 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 3
Dizziness (Nervous system disorders) | 0 | 3 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 4 | 4 | 1 | 3 | 1
Hypertension (Vascular disorders) | 1 | 1 | 2 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.